CLINICAL TRIAL: NCT03577392
Title: Effect of Intravenous Pump of Recombinant Human Endostatin Combined With XELOX Chemotherapy, and a Potential Prognostic Biomarkers in Patient With Advanced Colorectal Cancer
Brief Title: Recombinant Human Endostatin in Combination With XELOX Therapy in Patient With Advanced Colorectal Cancer.
Acronym: EXECC
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Collaborators: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, ming zeng, MD, Director of Cancer Center, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SIM-ED-1512
Record Dates: First submitted 2018-06-23; First posted 2018-07-05 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Quality of Life
MeSH Terms: interventions — Oxaliplatin; Capecitabine

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to receive either three treatment cycles of intravenous pump of recombinant human endostatin before chemotherapy.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XELOX chemotherapy with recombinant human endotatin (Experimental): Patients received a triweekly treatment cycle.Oxaliplatin(130mg/m2 over 2h)was intravenously administated for at least 2h on day 1. Capecitabine(1000mg/m2 twice daily)was oral administrated from the evening of day 1 to the morning of day 15.The dose of Recombinant human endostatin on day -5 was calculated according to the patients's body surface area, to provide a CIV 7 days' dose in physiological saline to 240mL volume.
  Interventions: Drug: oxaliplatin + capecitabine (XELOX chemotherapy); Drug: rebombniant human endostatin
- XELOX chemotherapy without recombinant human endotatin (Active Comparator): Patients received a triweekly treatment cycle.Oxaliplatin(130mg/m2 over 2h)was intravenously administated for at least 2h on day 1. Capecitabine(1000mg/m2 twice daily)was oral administrated from the evening of day 1 to the morning of day 15.
  Interventions: Drug: oxaliplatin + capecitabine (XELOX chemotherapy)

INTERVENTIONS:
Drug: oxaliplatin + capecitabine (XELOX chemotherapy) — Oxaliplatin(130mg/m2 over 2h)was intravenously administated for at least 2h on day 1. Capecitabine(1000mg/m2 twice daily)was oral administrated from the evening of day 1 to the morning of day 15.
Drug: rebombniant human endostatin — Endostar is a recombinat human endostatin with antiangiogenic properties that has been useful in treating a wide range of cancers and shows promise for use in combination treatment for advanced colorectal cancer. The dose of Recombinant human endostatin on day -5 was calculated according to the patients's body surface area, to provide a CIV 7 days' dose in physiological saline to 240mL volume.
  Arms: XELOX chemotherapy with recombinant human endotatin

SUMMARY:
To study safety and efficacy of intravenous pump of recombinant human endostatin combined with XELOX-treated and also investigate the potential value of CECs level for the prediction of PD and outcomes in patients with advanced colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Clear pathology diagnosis of stage for the Ⅳ period of advanced colorectal cancer.
* There are at least 1 imaging examinations according to the standard of RECIST（the longest diameter is at least 10mm with spiral CT and 20mm with ordinary CT）.
* Male or female , age 18～75
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* The patients had to have a life expectancy of at least 3 months.
* A white blood count (WBC) greater than 3000/mm3, platelets greater than 100 000/mm3, and normal coagulation values.
* Aspartate aminotransferase (AST) and adenosine triphosphate (ALT) values were to be less than 2.5 times the upper limit of normal;a bilirubin level of less than 25 lmol/l；a creatinine value less than 130 lmol/l.
* Informed consent was obtained from all patients.

Exclusion Criteria:

* Patients having a brain tumor or brain metastases, a bleeding disorder, receiving anti-coagulant therapy.
* a history of myocardial infarction or angina pectoris in the last 6 months or uncontrolled congestive heart failure, having an active infection or receiving radio- or chemotherapy within 4 weeks before study.
* patients with uncontrolled serious medical or psychiatric illness or having any other condition that was likely to interfere with regular follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 4 years
  Evaluate the effect of XELOX therapy with or without recombinant human endostatin on progression free survival

SECONDARY OUTCOMES:
local control | 4 years
  To describe local control and out-of-field disease progression
Overall survival | 4 years
  comparison to maintenance XELOX chemotherapy alone.

CONTACTS AND LOCATIONS:
Overall Officials: Ke Xie, MD PhD, Study Chair — Sichuan Provincial People Hospital
Locations (1):
- Sichuan Provincial People Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No